CLINICAL TRIAL: NCT05664191
Title: Use of Levosimendan as Treatment of Aneurysmal SubArachnoid Hemorrhage
Brief Title: Levosimendan as Treatment of Aneurysmal SubArachnoid Haemorrhage
Acronym: LEVOSAH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP200175
Record Dates: First submitted 2022-07-28; First posted 2022-12-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Sub-arachnoid Haemorrhage
Keywords: Sub-arachnoid haemorrhage; vasospasm; delayed cerebral ischemia; stroke
MeSH Terms: conditions — Stroke | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LEVOSIMENDAN (Experimental): Experimental : Levosimendan group
  Interventions: Drug: Levosimendan
- PLACEBO (Placebo Comparator): Placebo : Comparator group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levosimendan — Infusion at 0.1 µg/kg/min at day 1 and day 8
  Arms: LEVOSIMENDAN
Other: Placebo — Glucose 5%, solution for injection ECOFLAC at day 1 and day 8
  Arms: PLACEBO

SUMMARY:
Sub-arachnoid haemorrhage (SAH) are often due to ruptured intracerebral aneurysms and are associated with an importante morbi-mortality. SAH are often complicated by delayed cerebral ischemia (DCI) potentially due to cerebral vasospasm (CVS). A recent study showed that levosimendan, an inotropic and vasodilatory drug, could reduce the incidence of CVS and potentially improve patient outcome.

In this pilot randomized controlled trial, we will evaluate the impact Levosimendan vs Placebo in SAH patient on the occurrence of CVS and DCI.

Study population: adult patient admitted to ICU for aneurysmal SAH WFNS grade I-IV and mFisher 3-4.

Intervention: Levosimendan (0.1 µg/kg/min) or placebo infusion at Day 1 and 8.

Primary outcome: incidence of DCI or CVS at day 14

Duration of the study: 24 months

Number of patients: 30 (15 patients per group) Number of center: 1

DETAILED DESCRIPTION:
Background

Aneurysmal subarachnoid hemorrhage (aSAH) is a frequent type of stroke. It is associated with a significant morbidity and mortality and particularly affects young subjects. Complications that can occur after an aSAH include acute cardiac dysfunction and cerebral arterial vasospasm (CVS), which produces delayed cerebral ischemia (DCI). These complications are associated with a worsened outcome for aSAH patients. There is no proven preventive treatment for these complications.

Clinical and experimental data show that Levosimendan could be ideal to prevent these complications. In a recent study (Trinh-Duc et al, Crit Care 2021), treatment with Levosimendan was associated with a reduced incidence of CVS in a SAH patients.

The use of levosimendan, a non-catecholaminergic vasodilator inotrope in a context of already maximal endogenous adrenergic stimulation, thus seems to be suitable and able to improve the prognosis of aSAH patients.

Experimental design

Single-center, phase II, comparative, randomized, superiority, placebo-controlled, double-blind, pilot drug trial using Bayesian inference.

Study drug

Patient treated with levosimendan infusion at 0.1 microgram/kg/min for 24 hours at D1 and D8.

Number of patients

30 patients, i.e. 15 patients per group

Number of centre : 1

Duration of inclusion: 24 months

Total duration of the trial: 27 months

Statistical analysis

Primary endpoint:

The proportion of patients with at least one of the following: death, vasopasm, or DCI within 14 days of inclusion will be compared using Bayesian analysis.

Secondary endpoints:

* Qualitative secondary endpoints will be analyzed by Chi-2 test. An exact probability test will be used if the Chi-2 validity criteria are not met.
* Quantitative secondary endpoints will be compared by Student's t test. Qualitative secondary endpoints will be compared by Wilcoxon test
* The evolution of mortality will be compared using a log-rank test
* The tests will be two-sided at the 5% significance level.

Support

This study is supported by Assistance Publique - Hôpitaux de Paris (AP-HP) and Orion Pharma.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (18 to 75 years old),
* hospitalized in surgical intensive care at Lariboisière Hospital for subarachnoid haemorrhage of aneurysmal origin
* WFNS clinical score of I to IV and a mFisher score of 3 or 4.

Exclusion Criteria:

* pregnant women
* contraindications to levosimendan (including hypersensitivity to levosimendan, severe hypotension (mean arterial pressure less than 65 mmHg), tachycardia (heart rate greater than 120 bpm), cardiac mechanical obstructions)
* severe renal failure (creatinine clearance < 30 ml/min)
* severe hepatic failure (signs of hepatic encephalopathy) or chronic liver disease
* history of torsades de pointes
* pre-existing severe neurovascular pathologies.
* Moribund patients.
* Patient not affiliated to social security
* Patient participating in another interventional research
* Patients under legal guardianship or curatorship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
SAFETY / TOLERABILITY / EFFICACY | within 14 days of inclusion
  Proportion of patients with at least one of the following: death, vasopasm, or DCI within 14 days of inclusion.
SAFETY / TOLERABILITY / EFFICACY | day 14, day 28, day 90
  Cumulative incidence of mortality, DCI, and vasospasm mRS score at 3 months Value of peak serum catecholamines (norepinephrine, adrenaline) within 5 days of admission Number of days alive at D14 without catecholamines and maximum dose (norepinephrine, dobutamine, dopamine, adrenaline, isoprenaline) if used.
  Time to peak troponin and BNP and their values Systolic and diastolic heart function assessed by echocardiography Daily clinical evolution with Glasgow score Daily transcranial doppler evolution Occurrence and extent of secondary cerebral ischemia diagnosed by systematic MRI at 3 months.
  Length of stay in the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Glen Chousterman, Study Director — Hôpital Lariboisière
Locations (1):
- Hôpital Lariboisière, Service d'anesthésie Réanimation, Paris, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trinh-Duc A, Labeyrie MA, Caillard A, Ben Hassen W, Mebazaa A, Chousterman BG. Effects of levosimendan on occurrence of cerebral vasospasm after aneurysmal subarachnoid hemorrhage: a case-control study. Crit Care. 2021 Nov 16;25(1):396. doi: 10.1186/s13054-021-03824-x. No abstract available. PMID 34784938